CLINICAL TRIAL: NCT02147743
Title: Preventing Adolescents From Entering the Juvenile Justice System: Testing An Empirically-Supported, Family-Based Diversion Model
Brief Title: Preventing Adolescents From Entering the Juvenile Justice System
Acronym: CCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Howard Liddle, Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 20080174
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Substance Use; Delinquency
Keywords: Adolescents; Family-Based treatment; Multidimensional Family Therapy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCP+MDFT (Experimental): Multidimensional Family Therapy (MDFT) is a multisystemic, flexible intervention system (Liddle, 2002). It is a strengths-based approach promoting protective factors and reducing risk factors for delinquency, substance use, and school problems. MDFT organizes interventions in key areas of the teen's life: self of the adolescent (includes HIV-STD risk behaviors), parenting, family environment, and school/vocational functioning.
  Interventions: Behavioral: CCP+MDFT
- CCP+SAU (Other): Services as Usual (SAU) are determined on a case-by-case basis by the CCP Case Manager. SAU includes a variety of services offered by a number of community partners.
  Interventions: Behavioral: CCP+SAU

INTERVENTIONS:
Behavioral: CCP+MDFT — Multidimensional Family Therapy (MDFT; Liddle, 2002) is one of a new generation of multi-systems oriented family-based intervention for adolescent substance abuse and delinquency. It has demonstrated considerable success with juvenile justice youth at various stages of their involvement in the justice system. The model has demonstrated efficacy in reducing substance use and delinquency, increasing the prosocial behaviors (e.g., family functioning, school outcomes) of substance abusing and court involved adolescents.
  Arms: CCP+MDFT
Behavioral: CCP+SAU — Services As Usual community partners will provide individualized mental health counseling and psychiatric services, psychoeducational groups and substance abuse counseling.
  Arms: CCP+SAU

SUMMARY:
This randomized controlled study tests an innovative juvenile diversion model that integrates evidence-based family therapy.Immediate and longer term effects of the family intervention will be compared to Services As Usual with 120 adolescents participating in Miami-Dade's Civil Citation Program.

DETAILED DESCRIPTION:
This study proposes to rigorously test the innovative Civil Citation Program (CCP)with an integrated evidence-based family intervention, Multidimensional Family Therapy[MDFT](Liddle, 2002).

The study sample includes youth referred to the CCP throughout Miami-Dade county and who according to CCP screening are rated as high risk for re-offending. Youth are 12-17 years old with a first or second misdemeanor charge (excluding any gang, violence, or sex crimes charge). Nearly all (97%) of these youth are ethnic minorities (Hispanic and African American). They are at risk for school failure, substance use, and chronic delinquency due to drug availability in their communities, poor family functioning, peer drug use/delinquency, and school failure / disengagement.

120 youth who enter the Civil Citation Program and are eligible for the study will be assigned to one of the two interventions: CCP+SAU or the experimental intervention, CCP+MDFT.

The study asks a classical services research question(Compton et al, 2005) - does the addition of a family therapy intervention, multidimensional family therapy, into an existing diversion program significantly enhance the program outcomes in key outcome domains: recidivism, substance use, delinquency, school and family functioning.

ELIGIBILITY:
Inclusion Criteria:

* Youth 12 to 17 years old
* Parent or guardian willing to participate in assessments/treatment
* Demonstrate risk for mental health, substance abuse, or anger/adjustment problems on the Juvenile Services Department screening warranting intervention but not requiring residential treatment

Exclusion Criteria:

* Youth under the age of 12 or over the age of 18
* Parent/guardian not willing to participate in assessments and treatment
* Youth not demonstrating mental health, substance abuse or anger/adjustment problems
* Youth requiring residential treatment
* Youth with severe mental illness or retardation

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Delinquency | Intake through 9-month follow-up
  Youth in CCP+MDFT will show less delinquency from intake to 9 months than youth in CCP+SAU.
  National Youth Survey Self-Report Delinquency Scale (SRD)will be used to assess delinquency.
Recidivism | 6 months prior to arrest that got youth in the CCP through 24 months after the baseline assessment
  Juvenile justice arrest records recoding total arrests, total misdemeanor arrests, and total felony arrests for youth 6 months prior to baseline through 24 months after baseline.

SECONDARY OUTCOMES:
Substance Use | Intake through the 9-month follow-up
  Youth in CCP+MDFT will report less substance use from intake to 9 months than CCP+SAU. The Timeline Follow-Back Method, Personal Experiences Inventory and Urinalyses will be used to measure substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Liddle, EdD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States